CLINICAL TRIAL: NCT03536416
Title: Multifaceted Theory-based Self-management Intervention to Improve Adolescents' Asthma Control: A Cluster-randomised Controlled Trial (RCT)
Brief Title: Self-management Intervention to Improve Adolescents' Asthma Control
Acronym: MAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Jonathan Grigg, Professor, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MGU0400
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Asthma
Keywords: Self-management; Children and young people; Schools
MeSH Terms: conditions — Asthma | interventions — Schools

STUDY DESIGN:
Intervention Model Description: The study will include three treatment arms. The first arm will receive the theatre workshop only; the second arm will receive the theatre workshop and the self-management workshops; the control group will receive usual care. Schools will be randomised to one of the groups.
Who Masked: Participant
Masking Description: The schools will be randomised, and will not be told which group they have been randomised to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Asthma workshop and theatre group (Experimental): My Asthma in School. This group will receive the self-management workshops for asthmatic children and the theatre performance for the whole year group.
  Interventions: Behavioral: My Asthma in School
- Theatre only group (Active Comparator): My Asthma in School. This group will receive the theatre performance only.
  Interventions: Behavioral: My Asthma in School
- Control group (No Intervention): My Asthma in School. The control group will receive usual care for the duration of the intervention.

INTERVENTIONS:
Behavioral: My Asthma in School — The intervention will include three arms. During the theatre workshop, the children will watch a theatre performance, and engage in a discussion at the end of the play, about what they have watched. The self-management workshops will cover a range of topics identified as barriers to self-management in our earlier study, and will be delivered to children with asthma only. The control group will receive usual care during the intervention.
  Arms: Asthma workshop and theatre group; Theatre only group

SUMMARY:
Approximately 1.1 million children and young people in the United Kingdom (UK) are living with asthma, making it the most common chronic disease in children in the UK. Our recent observational study found that poor asthma control, poor medication adherence, and a poor understanding of asthma were key unmet needs of secondary school children. Following the findings from an earlier study, the investigators have developed a preliminary theory-based multi-faceted intervention, aimed at improving asthma self-management and control in young people.

DETAILED DESCRIPTION:
The investigators have developed a theory-driven self-management intervention for children and young people which addresses the barriers to successful self-management, which were identified in an earlier study. The intervention will engage asthmatic teenagers and their peers, and will be delivered in two components. The first component includes a theatre workshop for all children aged 11-13 years in London secondary schools. The aim of this component is to raise awareness of asthma in schools among peers. The second component is a series of four self-management workshops for children with asthma. The aim of this component is to teach children about asthma, using interactive role plays and games. The main topics will include asthma general knowledge and understanding; General Practitioner (GP) communication; asthma triggers and symptoms; medication and emergency response; and self-management techniques and goal setting. The children will also receive a toolkit to take home with them, which will include a copy of the workbook that they have used during the day, containing information on what they have learnt. There will also be information on where they can get more help for their asthma. The toolkit will also include information about a smartphone gaming app, which will be about asthma knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Doctor-diagnosed asthma
* Aged 11-14 years (UK school years 7-8)
* Attending the secondary school in which the study is implemented
* All children in years 7 and 8 in UK secondary schools are eligible to watch the theatre performance

Exclusion Criteria:

* No diagnosis of asthma
* Not aged 11-14 years (UK school years 7-8)
* Not attending the school at the time the intervention is delivered

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Asthma control | 15 months
  This will be measured using the validated Asthma Control Test. Scores range from 5-25. A score of 19 or below indicates poorly controlled asthma; a score of 20 or above indicates good asthma control.

SECONDARY OUTCOMES:
Medication Adherence Rating Scale. | 15 months
  Measures medication adherence. This scale includes 10 questions. Compliance is indicated by a 'no' response to questions 1-6 and 9-10, and a 'yes' response for questions 7 and 8.
Unscheduled care | 15 months
  This scale includes two multiple choice questions; one about unplanned doctor visits and one about unplanned hospital emergency department visits over the previous four weeks.
Brief-Illness Perception Questionnaire | 15 months
  This scale includes 9 questions about perceptions of illness. Questions 3, 4 and 7 are reverse scored, and added to the scores for the remaining questions. A higher score indicates a more threatening view of the illness.
School absences | 15 months
  This scale includes 3 multiple choice questions. These questions measure whole school day absences, lesson absences, and Physical Education lesson absences, over a four-week period.
Asthma knowledge | 15 months
  This scale includes 14 questions about asthma knowledge.
Beliefs About Medicines Questionnaire | 15 months
  This scale includes 10 statements about asthma medication. The participants indicate their agreement with the statement by selecting an option from strongly agree to strongly disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Overall findings for each school will be reported back to individual schools, however individual participant data will not be reported due to data protection and confidentiality.

REFERENCES:
- [Background] Mosler G, Harris K, Grigg J, Steed L. Developing a theory-based multimedia intervention for schools to improve young people's asthma: my asthma in school (MAIS). Pilot Feasibility Stud. 2020 Sep 2;6:122. doi: 10.1186/s40814-020-00670-6. eCollection 2020. PMID 32884832
- [Background] Harris K, Mosler G, Grigg J. Theory-based self-management intervention to improve adolescents' asthma control: a cluster randomised controlled trial protocol. BMJ Open. 2019 Apr 23;9(4):e025867. doi: 10.1136/bmjopen-2018-025867. PMID 31015270
- [Background] Mosler G, Euba T. Taking control through drama. Lancet. 2018 Jan 27;391(10118):303-304. doi: 10.1016/S0140-6736(17)32283-3. Epub 2017 Sep 8. No abstract available. PMID 29413036
- [Result] Harris K, Newby C, Mosler G, Steed L, Griffiths C, Grigg J. School-based self-management intervention using theatre to improve asthma control in adolescents: a pilot cluster-randomised controlled trial. Pilot Feasibility Stud. 2022 Mar 23;8(1):67. doi: 10.1186/s40814-022-01031-1. PMID 35321754
- See also: Project website — https://myhealthinschool.org/